CLINICAL TRIAL: NCT06657664
Title: Effect of Cryotherapy and Laser on Post-Operative Pain in Single Visit Endodontically Treated Symptomatic Apical Periodontitis Cases
Brief Title: Effect of Cryotherapy and Laser Application on Post-Operative Pain in Single Visit Endodontically Treated Symptomatic Apical Periodontitis Cases
Acronym: LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rawda Nashy, Rawda Nashy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TantaU 55
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Irriversible Pulpitis With Apical Peridontitis; Hot Tooth
Keywords: cryotherapy Low Level Laser Therapy LLLT single visit endodontic treatment irriversible pulpitis Apical peridontitis
MeSH Terms: interventions — Cryotherapy; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical study.
Masking Description: all participants have an equal chance to be enrolled in any of the study groups. This pattern was the most suitable way to ensure the balance of the anonymous prognostic factors in the participants between the three groups thus, eliminating the selection or allocation bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- control Group (Active Comparator): all occlusal contacts are reduced by 1 mm
  Interventions: Procedure: Control (Standard treatment)
- intracanal cryotherapy (Active Comparator): the root canals are given a final irrigation with 20 mL cold (2.5oC) saline solution for 5 minutes
  Interventions: Procedure: cryotherapy with sterile saline at 2.5ºC
- intraoral cryotherapy group (Active Comparator): ice sticks (wrapped in sterile gauze if needed) using plastic pipette droppers filled with freezing sterile water are placed intraorally in the mouth on the apices of the treated tooth on both buccal and palatal sides for 30 minutes
  Interventions: Procedure: intaoral cryotherapy
- Both intracanal and intraoral cryotherapy (Active Comparator): the root canals are given a final irrigation with 20 mL cold (2.5oC) saline solution for 5 minutes , the canal is obturated and then ice sticks (wrapped in sterile gauze if needed) using plastic pipette droppers filled with freezing sterile water are placed intraorally in the mouth on the apices of the treated tooth on both buccal and palatal sides for 30 minutes.
  Interventions: Procedure: Both intracanal and intraoral cryotherapy
- Low Level Laser Therapy (Active Comparator): laser irradiation on the soft tissues covering the apices of the tooth on both buccal and palatal surfaces respectively.
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Procedure: cryotherapy with sterile saline at 2.5ºC — the root canals are given a final irrigation with 20 mL cold (2.5oC) saline solution for 5 minutes before obturation
  Other Names: iced intracanal saline; intracanal cryotherapy
  Arms: intracanal cryotherapy
Procedure: intaoral cryotherapy — ice sticks (wrapped in sterile gauze if needed) using plastic pipette droppers filled with freezed sterile water are placed intraorally in the mouth on the apices of the treated tooth on both buccal and palatal sides for 30 minutes
  Arms: intraoral cryotherapy group
Procedure: Both intracanal and intraoral cryotherapy — Canal is irrigated with iced saline for 5 minutes before obturation . Root canal is obturated and coronal restoration is done. Then, application of intraoral cryotherapy is performed by ice sticks for 30 minutes.
  Arms: Both intracanal and intraoral cryotherapy
Device: Low Level Laser Therapy — laser irradiation on the soft tissues covering the apices of the tooth on both buccal and palatal surfaces respectively
  Other Names: photobiomodulation; LLLT; cold lasers
  Arms: Low Level Laser Therapy
Procedure: Control (Standard treatment) — , all occlusal contacts were reduced by 1 mm
  Other Names: occlusal reduction
  Arms: control Group

SUMMARY:
This study compare the effect of applying ice after single visit endodontic treatment with lasers to reduce post operative pain .

DETAILED DESCRIPTION:
one of the most popular complications after single visit endodontic treatment is pain either spontaneous or on biting so in this study we choose one of the most difficult and challenging cases " Hot tooth " to compare lasers and cryotherapy different applications to reduce post operative pain after single visit endodontic treatment

ELIGIBILITY:
Inclusion Criteria:

* • Vital teeth display symptomatic apical periodontitis (Symptomatic apical periodontitis was determined based on the clinical symptoms of severe preoperative pain (visual analogue scale [VAS] > 60) and severe percussion pain (VAS > 60).

  * Teeth, with a periapical index score (PAI) of 2 or 3 indicating small changes in bone structure and slight mineral loss respectively.
  * Mobility less than 1 mm in either direction.
  * Absence of periodontal pocket around the tooth.
  * Symptomatic pulpitis with spontaneous pain or lingered by cold or heat.
  * Teeth without pus or inflammatory exudates draining through the canal.
  * Teeth without anatomic variations

Exclusion Criteria:

* • Patient with any systemic disease.

  * Immunocompromised patients.
  * Pregnant or lactating patients.
  * Apparently narrow roots in which apical preparation with the #40 file would be overzealous.
  * Retreatment cases.
  * Necrotic painful teeth with absence of sinus tract for drainage.
  * Patients on analgesics or sedative medication up to 6 hours before treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
post operative pain | preoperative, after 24 hours, on the third , fifth, one week & two weeks after treatment
  post operative pain and pain on percussion is tested using visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided